CLINICAL TRIAL: NCT06361966
Title: Evaluating User Satisfaction and Feasibility of a Remote-digital Model for 3d Scanning and Printing of Prosthetic Sockets for Patients With Transtibial Amputation: A Preliminary Clinical Trial
Brief Title: Evaluating User Satisfaction and Feasibility of a Remote Model for 3d Scanned and Printed Transtibial Prosthetic Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Prosfit Technologies JSC (Unknown); Centre for Allied Health and Pharmacy Excellence (CAPE) (Unknown)
Responsible Party: Principal Investigator, Tabitha Quake, Principal Prosthetist/Orthotist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021/00638
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Amputation; Prosthesis User
Keywords: transtibial amputation; transtibial prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminate socket (Active Comparator): control intervention as standard treatment for transtibial amputees requiring a lower limb prosthesis
  Interventions: Device: 3d printed prosthetic socket
- 3d printed socket (Experimental): trial intervention for transtibial amputees requiring a lower limb prosthesis
  Interventions: Device: 3d printed prosthetic socket

INTERVENTIONS:
Device: 3d printed prosthetic socket — 3d printed prosthetic socket produced through multi-jet fusion (MJF)

SUMMARY:
The goal of this clinical trial is to investigate the repeatability of application of a fully remote method of manufacturing 3D printing of prosthetic sockets for transtibial amputees, and determine user satisfaction of sockets produced through these methods. The study also aims to evaluate the time and cost effectiveness of this production model.

The main question[s] it aims to answer are:

1. To determine the repeatability and user satisfaction with transtibial sockets produced using a remote-digital method as compared to conventional manufacturing methods.
2. To determine if transtibial prosthetic users have greater prosthetic satisfaction scores across the 4 Prosthesis Evaluation Questionnaire (PEQ) subscales of Utility (UT), Appearance (AP), Sounds (SO) and Residual Limb Health (RL) with the 3D printed socket fabricated through the remote-digital method compared to the laminate socket made using the conventional method.
3. To determine if transtibial prosthetic users experience greater socket comfort with the 3D printed socket compared to the laminate socket.

Participants will receive a 3D printed socket (trial intervention) and a laminate socket (control intervention) and will use each socket for a period of 4 weeks.The order of socket use will be randomised. At the end of each 4 week period, participants will rate their comfort and satisfaction with the socket. At the end of the trial, participants will indicate their preferred socket, which will be fitted to their prosthesis.

Participants will attend 6 visits across a total duration of 11 weeks during the course of the study.

DETAILED DESCRIPTION:
The visit schedule for the study is as follows:

* Visit 1 (Week 0): Attain consent and initiate casting and scanning process for 1 laminate and 1 3D printed transtibial socket
* Visit 2 (Week 3): Fitting and adjustment of first prosthetic socket (either 3D printed or laminate socket). Subjects to rate comfort of first socket.
* Visit 3 (Week 5): Follow-up on any required device adjustments/ troubleshooting to first socket.
* Visit 4 (Week 7): Evaluation of user satisfaction with first socket. Subjects to fill up survey on first socket. Fitting of other socket design (second socket). Subjects to rate comfort of second socket.
* Visit 5 (Week 9): Follow-up on any required device adjustments/ troubleshooting to second socket.
* Visit 6 (Week 11): Evaluation of user satisfaction with second socket. Subjects to fill up survey on second socket and select their preferred socket. Fitting of patient's preferred socket to prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation, current transtibial prosthetic users minimally capable of community ambulation (mobility grades K2 - K4) who have completed gait training, current users of a roll on elastomeric or silicone liner system, and aged 21 years old and above to be able to provide informed consent.

Exclusion Criteria:

1. Functional status: patients with severe aphasia or neglect (inability to obey 1 step commands), communication disorders precluding understanding of instructions, cognitive impairment, dementia, untreated depression or psychiatric disorder.
2. Mobility status: patients who are non-community ambulators (mobility grade K1) or who have not completed gait training
3. Active limb conditions: uncontrolled lower limb volume fluctuations, severe stump varus or valgus deformities and/or lower limb contractures of over 10 degrees, or with local limb conditions which could be exacerbated by research interventions such as open wounds, ulcers, stump pain or stump wounds/ulcers, neuromas, active arthritis or joint or limb pain.
4. Reproductive age females should not be pregnant during the study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Prosthesis Evaluation Questionnaire | after 4 weeks of socket use
  Subscales of Utility, Appearance, Sounds and Residual Limb Health, and an individual satisfaction question
Socket Comfort Score | at initial socket fitting and 4 weeks post-fitting
  Self-reported socket comfort is rated from 0 - 10, where 0 is the most uncomfortable socket imaginable and 10 the most comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Tabitha Quake, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No